CLINICAL TRIAL: NCT02234479
Title: A Pilot Study: Topical Application of Medihoney for Management of Radiation Dermatitis
Brief Title: MediHoney for Radiation Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Integra LifeSciences Corporation (Industry)
Responsible Party: Principal Investigator, Department of Radiation Oncology, Principle Investigator, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00058645
Record Dates: First submitted 2014-09-02; First posted 2014-09-09 (Estimated); Results first posted 2016-08-08 (Estimated); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Breast Cancer; Radiation Dermatitis
Keywords: Breast Cancer; Radiation Dermatitis
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hydrophor (Group A) (Active Comparator): Group A (current standard of care): Patients will be instructed (by nurses and with printed study materials) to apply a thin layer of the Hydrophor daily, starting at the onset of radiation therapy (RT) and continuing until 2 weeks after the final RT session or until the RT site is healed (whichever is first). Hydrophor application should include the entire treatment area, including the axillae and shoulder/back area in patients treated with modified radical mastectomy. To avoid possible build-up effects, patients should not apply the Hydrophor within 4 hours of receiving RT. Patients should wash the application area daily with perfume-free soap and tap water. Patients will be asked to refrain from using other topical agents in the irradiated area.
  Interventions: Biological: Hydrophor (Group A)
- MediHoney (Group B) (Experimental): Group B (study target): Patients will be instructed (by nurses and with printed study materials) to apply a thin layer of the Medihoney daily, starting at the onset of RT and continuing until 2 weeks after the final RT session or until the RT site is healed (whichever is first). Medihoney application should include the entire treatment area, including the axillae and shoulder/back area in patients treated with modified radical mastectomy. To avoid possible build-up effects, patients should not apply the Medihoney within 4 hours of receiving RT. Patients should wash the application area daily with perfume-free soap and tap water. Patients will be asked to refrain from using other topical agents in the irradiated area.
  Interventions: Biological: MediHoney (Group B)

INTERVENTIONS:
Biological: Hydrophor (Group A) — * Rehydrates dry, chapped or chafed skin
  * May be used alone as a skin lubricant or protectant
  Arms: Hydrophor (Group A)
Biological: MediHoney (Group B) — It helps the body's natural healing processes in three key ways which have been shown to have healing benefits:
  * Maintain a balanced environment for healing.
  * Aids in reducing dermatitis.
  * Reduce affected area pH.2-3
  Arms: MediHoney (Group B)

SUMMARY:
The aim of this study is to compare the effects of Medihoney and Hydrophor on radiation dermatitis reactions in a group of women undergoing radiation therapy for breast cancer. It is hoped that the outcome of this pilot study will provide evidence supporting the use of Medihoney in preventing and treating radiation dermatitis as well as sufficient preliminary data to expand this study to larger, federally funded research (R01) looking at the beneficial aspects of Medihoney across a spectrum of radiation dermatitis and mucositis in several disease settings.

DETAILED DESCRIPTION:
Background: Radiation dermatitis, also known as radiodermatitis or radiation skin reaction, is a widely reported side effect of radiation therapy in cancer. The most common radiation therapy-induced side effect is acute skin reaction, which can range from mild erythema to confluent moist desquamation. Almost all patients receiving radiation therapy have a risk of developing radiation dermatitis (Trueman, 2012).

When not managed appropriately, radiation dermatitis can affect patients' physical functioning and quality of life. It can also cause pain and discomfort and may result in infection and/or interruption of treatment (Feight et al., 2011). An important role for oncology nurses is in educating, assessing, and monitoring patients for radiation dermatitis. Many nursing interventions are in use, including those based on tradition, physician preference, and published reports. In routine practice, most interventions for radiation dermatitis are institution-specific and not reliably evidence based.

At the investigators institution, Hydrophor (Aquaphor), an ointment containing petrolatum, mineral oil, ceresin, and lanolin alcohol is the current standard of care for preventing and treating radiation dermatitis. Some women under treatment for breast cancer report disliking the smell and/or texture of Hydrophor. Rarely reported side effects have included allergic reactions, burning, stinging, and/or redness. Honey is an ancient remedy that has most recently shown promising results in treating burns, oral infections, and promoting surgical wound healing and palliation. The topical application of honey has been reported to be advantageous in radiation mucositis (Biswal et al., 2003). In a continuing effort to identify those treatment options that can make the investigators patients more comfortable and reduce complications from radiation dermatitis, the investigators are interested in conducting a small pilot study comparing the effectiveness of a honey-based treatment (Medihoney) with that of the investigators current standard of care (Hydrophor).

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer treated with either lumpectomy or mastectomy (with or without reconstruction).
* The patient must be female.
* Radiation therapy planned to whole breast/chestwall area (can include lymph node radiation; conventional 3D radiation, IMRT/IGRT, and hypofractionation are all allowed).
* Age ≥ 18 years old.

Exclusion Criteria:

* Previous radiation therapy to chest area that would result in overlapping radiation fields.
* Wound care issues.
* Patients undergoing concurrent cytotoxic chemotherapy and radiation therapy (concurrent Herceptin and/or tamoxifen/aromatase inhibitors and RT is allowed).
* Patients receiving HDR (savi or mammosite) brachytherapy treatments.
* Patients with an allergy and/or sensitivity to Hydrophor, honey, and/or Medihoney.
* Immunocompromised status.
* Age < 18 years old.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2014-06; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Nichols, MD, Principal Investigator — University of Maryland, College Park
Locations (1):
- University of Maryland, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Hydrophor (Group A): Group A (current standard of care): Patients will be instructed (by nurses and with printed study materials) to apply a thin layer of the Hydrophor daily, starting at the onset of radiation therapy (RT) and continuing until 2 weeks after the final RT session or until the RT site is healed (whichever is first). Hydrophor application should include the entire treatment area, including the axillae and shoulder/back area in patients treated with modified radical mastectomy. To avoid possible build-up effects, patients should not apply the Hydrophor within 4 hours of receiving RT. Patients should wash the application area daily with perfume-free soap and tap water. Patients will be asked to refrain from using other topical agents in the irradiated area.
  Hydrophor (Group A): •Rehydrates dry, chapped or chafed skin
  •May be used alone as a skin lubricant or protectant
- MediHoney (Group B): Group B (study target): Patients will be instructed (by nurses and with printed study materials) to apply a thin layer of the Medihoney daily, starting at the onset of RT and continuing until 2 weeks after the final RT session or until the RT site is healed (whichever is first). Medihoney application should include the entire treatment area, including the axillae and shoulder/back area in patients treated with modified radical mastectomy. To avoid possible build-up effects, patients should not apply the Medihoney within 4 hours of receiving RT. Patients should wash the application area daily with perfume-free soap and tap water. Patients will be asked to refrain from using other topical agents in the irradiated area.
  MediHoney (Group B): It helps the body's natural healing processes in three key ways which have been shown to have healing benefits:
  * Maintain a balanced environment for healing.
  * Aids in reducing dermatitis.
  * Reduce affected area pH.2-3
Period: Overall Study
Arm/Group | Hydrophor (Group A) | MediHoney (Group B)
Started | 16 | 18
Completed | 15 | 15
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hydrophor (Group A) | MediHoney (Group B) | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 40 [18 to 75] | 40 [18 to 75] | 40 [18 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 18 | 34
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 7 | 10
  White | 13 | 11 | 24
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Whom Received Medihoney Treatment and Were Analyzed Weekly for Skin Changes While Undergoing Radiation Therapy
Description: The aim of this study is to compare the effects of Medihoney and Hydrophor on radiation dermatitis reactions in a group of women undergoing radiation therapy for breast cancer. It is hoped that the outcome of this pilot study will provide evidence supporting the use of Medihoney in preventing and treating radiation dermatitis as well as sufficient preliminary data to expand this study to larger, federally funded research (R01) looking at the beneficial aspects of Medihoney across a spectrum of radiation dermatitis and mucositis in several disease settings.
Time Frame: 12 months
Population: Participants were analyzed for skin changes (during weekly visits with physician) during radiation treatment. Only 15 participants from each group completed the study, 1 subject from Group A and 3 subjects from Group B withdrew.
Measure: Number; unit: participants
Arm/Group | Hydrophor (Group A) | MediHoney (Group B)
Number analyzed (Participants) | 16 | 18
participants
  radiation dermatitis | 15 | 15
  hyperpigmentation | 15 | 15

ADVERSE EVENTS:
Time Frame: Adverse event data were collected in a 6 month period.
Arm/Group | Hydrophor (Group A) | MediHoney (Group B)
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 1/16 | 0/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrophor (Group A) (N=16) | MediHoney (Group B) (N=18)
dermatitis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No